CLINICAL TRIAL: NCT04426591
Title: Kinetics of Donor Red Blood Cell Survival in Sickle Cell Disease
Brief Title: Red Blood Cell Survival in Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Marianne Yee (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cerus Corporation (Industry)
Responsible Party: Sponsor-Investigator, Marianne Yee, Associate Professor, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00117580; 1K23HL146904 (NIH)
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease
Keywords: Chronic transfusion therapy
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Biotin labeled Red Blood Cells (Experimental): Participants receiving a transfusion with biotin labeled RBCs. Samples will be taken for 12 weeks after the biotinylated transfusion. During this time participants will continue to receive regular monthly transfusions (non-biotinylated) as part of CTT.
  Interventions: Drug: Biotin Labeled Red Blood Cells; Device: INTERCEPT Blood System

INTERVENTIONS:
Drug: Biotin Labeled Red Blood Cells — On the day of transfusion, a 20 mL aliquot will be sterilely withdrawn from each RBC unit, washed and labeled with sulfo-NHS-biotin for 30 minutes, washed to stop the labeling reaction, then resuspended in plasma to a hematocrit of ~60%. The biotin-labeled RBC (BioRBC) will be transfused along with the remainder of the RBC unit (unlabeled volume). Standard blood bank and CTT protocols and minor antigen matching for SCD patients will be followed. Exact transfusion volume will be determined based on pre-transfusion hemoglobin (Hb), sickle cell hemoglobin (HbS), and body weight, per clinical protocol.
Device: INTERCEPT Blood System — In addition to the blood drawn for the main study, individuals participating in this optional intervention will have additional tubes of peripheral venous blood will be drawn for evaluating treatment-emergent antibodies specific to INTERCEPT RBCs and acridine surface label monitoring. Tests for treatment-emergent antibodies specific to INTERCEPT RBCs will be performed according to procedures developed by Cerus Corporation.

SUMMARY:
This is a single-arm, mechanistic clinical trial to measure predictors of senescence and the in vivo survival of transfused red blood cells (RBCs) in individuals with sickle cell disease (SCD) receiving chronic transfusion therapy (CTT). Chronic transfusion in patients with SCD is a common treatment. The efficacy of RBC transfusion therapy to treat or prevent complications of SCD may be hampered by variable survival of the transfused donor RBC. The overall aim is to see how long RBC survive in SCD patients who are chronically transfused. When a study participant has a regular blood transfusion the researchers will label a small portion of the RBCs that are transfused with biotin. The participant will return at Day 1, weekly for 3 months and monthly for 3 months to measure how long those RBCs survive. An optional sub-study using INTERCEPT RBCs will mirror the main study but will use INTERCEPT RBCs that have biotinylated for 1 RBC unit.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) carries significant morbidity as a result of red blood cell (RBC) sickling and hemolysis. Stroke is one of the most devastating sequelae of SCD. Chronic transfusion therapy (CTT) reduces stroke risk by supplying normal, non-sickle RBC to circulation, thereby reducing the percentage of endogenous sickle RBC in circulation, and maintaining a higher hemoglobin (Hb), thereby suppressing erythropoiesis of new sickle RBC. While the efficacy of CTT in stroke prophylaxis is well-established, nearly 45% of children continue to have silent or overt strokes despite CTT. The failure of CTT to prevent stroke events may be related to inadequate reduction of circulating sickle RBC and erythropoiesis. The amount of circulating sickle-RBC is related to the survival kinetics of both transfused RBC and endogenous sickle RBC.

In a large, longitudinal analysis of CTT in SCD, the researchers found wide variation in the survival of donor RBC following transfusion, with faster clearance associated with patient immune features (historical RBC alloimmunization and spleen presence) and with donor RBC glucose-6-phosphate-dehydrogenase (G6PD) deficiency. To better understand the roles of patient and donor factors in the survival and clearance of transfused RBC, the researchers propose a mechanistic, clinical trial during chronic transfusion episodes in patients with SCD, in which a small aliquot of each transfused unit is labeled with biotin conjugated to RBC surface proteins, to safely identify and measure the in vivo survival of donor RBC.

Aim 1 will examine the relationships of the recipient's immune system (past alloimmunization, splenic volume, and markers of reticuloendothelial system function) on the post-transfusion survival of biotin-labeled donor RBC.

Aim 2 will examine the relationships of donor RBC G6PD levels and donor RBC metabolomics with the in vivo survival and changes in donor RBC senescence markers. Completion of these aims will increase the understanding of mechanisms for the variability in RBC survival during CTT, identifying donor and recipient risk factors for decreased RBC survival. Ultimately this knowledge will inform the management of CTT to improve the prevention of strokes in SCD.

Aim 3 will compare the in vivo survival and clearance rate of phenotype-matched RBCs prepared with an investigational pathogen-reduction system (INTERCEPT Blood System) vs. the in vivo survival and clearance rate of conventional, phenotype-matched RBCs (not treated with INTERCEPT). Biotin labeling of donor RBC will be used to measure RBC survival. This is an optional study activity for study participants.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobinopathy:

  * Any sickle cell disease genotype, or
  * Transfusion-dependent thalassemia (TDT)
* Receiving CTT for ≥3 months prior to enrollment.
* For participants with past BioRBC transfusion exposure, BioRBC antibody screens must have been conducted through at least 6 months post exposure, with negative results.

Exclusion Criteria:

* Anticipated cessation of CTT in the next ≤2 months
* Ongoing consumption of biotin or raw egg dietary supplements
* Antibody specific of INTERCEPT RBCs at baseline (for subjects consenting to the optional arm)
* BioRBC-specific antibodies ever detected in the past, or detected on post-enrollment screening prior to first infusion of Bio-RBC.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Number of Biotin Labeled RBCs | Day 1, Weeks 1-12
  Survival of the transfused biotin labeled RBCs will be assessed as the count of biotinylated RBCs per sample.
Half-life of Biotinylated RBCs | Up to Day 70
  Survival of transfused biotin labeled RBCs will be assessed as the half-life of biotinylated RBCs.
Mean Potential Lifespan (MPL) of Biotinylated RBCs | Up to Day 70
  The long-term lifespan of transfused biotin labeled RBCs is assessed as the linearly extrapolated as mean potential lifespan (MPL) of biotinylated RBCs.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Yee, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Hughes Spalding Children's Hospital, Atlanta, Georgia
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available for sharing with other researchers, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data will be made available for sharing immediately following publication, with no end date.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, for the purpose of achieving the aims in the approved proposal. Proposals should be directed to Marianne.Yee@choa.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04426591/ICF_000.pdf